CLINICAL TRIAL: NCT02927860
Title: Sleep and Activity Monitoring After Thoracic Surgery
Status: Terminated | Type: Observational
Why Stopped: Fitbit was not giving the necessary data.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mark Allen, Principal Investigator, Mayo Clinic
Other Study IDs: 16-006864
Record Dates: First submitted 2016-10-06; First posted 2016-10-07 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Thoracic Surgery; Surgery, Thoracic
Keywords: sleep; exercise; activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Fitbit — A FitBit HR monitor will be placed on patients when they arrive on the nursing unit after thoracic surgery. Sleep and activity will be monitored for the duration of the patient's hospitalization and the data from the Fitbit HR device will be downloaded by the study staff to a computer.

SUMMARY:
Show by collecting sleep and activity data, outcomes after thoracic surgery are improved with better sleep and increased activity.

DETAILED DESCRIPTION:
Little is known about how sleep deprivation affects recovery after thoracic surgery. There is some evidence that in cardiac surgery, sleep disturbance can lead to delayed recovery and mental status changes in the postoperative period. There are no similar reports of studies after thoracic surgery. We think that increased activity after surgery is beneficial for a rapid recovery and prevents blood clots, pneumonia and deconditioning. Without specific data this is difficult to prove.

ELIGIBILITY:
Inclusion Criteria:

* undergoing thoracic surgery at Mayo Clinic Rochester
* expected to stay in hospital for at least 4 days
* signed consent form

Exclusion Criteria:

* Unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mayo Clinic Rochester patients undergoing thoracic surgery
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2016-10; Primary Completion 2017-08-08 (Actual); Study Completion 2017-08-08 (Actual)

PRIMARY OUTCOMES:
Length of Stay | Until discharge, an average of 5 days

SECONDARY OUTCOMES:
Incidence of pneumonia while hospitalized | Until discharge, an average of 5 days
Incidence of blood clot while hospitalized | Until discharge, an average of 5 days
Incidence of deconditioning while hospitalized | Until discharge, an average of 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Allen, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No